CLINICAL TRIAL: NCT03607084
Title: Evaluating the Impact of School-based Health Programs on Children's Well-being and Academic Performance
Brief Title: School-based Health Programs on Children's Wellbeing in Lusaka, Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Healthy Kids/Brighter Future (Unknown)
Responsible Party: Principal Investigator, Günther Fink, Adjunct Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB15-1539
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Acute Disease; Morbidity
Keywords: school-aged children; school-based health program; Zambia; child and adolescent health
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group receives a school health program that has two components: the training of selected teachers to become school Health Workers and bi-annual health screenings of all students.
  Interventions: Behavioral: School Health Worker Program
- Control (No Intervention): The control group receives regular school programming.

INTERVENTIONS:
Behavioral: School Health Worker Program — The intervention trains selected teachers to deliver health lessons to students, perform basic first aid, recognize common illnesses, refer student to skilled medical attention when needed. The intervention provides schools with basic medical supplies including pain relief medication, thermometers, bandages, antiseptics, and oral rehydration solution. Vitamin A supplementation and presumptive deworming medication are administered to students during biannual health screenings.
  Arms: Intervention

SUMMARY:
This study evaluates the impact of a new and comprehensive school-based health program implemented in Lusaka, Zambia.

DETAILED DESCRIPTION:
While school-aged children in low- and middle-income countries remain highly exposed to acute infections, programs targeting this age group remain limited in scale and scope. In this study, we evaluate the impact of a new and comprehensive primary school-based health intervention program on student health outcomes and academic performance in Lusaka, Zambia. The intervention involved the training of teachers to become school health workers and the provision of vitamin A supplementation and deworming medication on a bi-annual basis. Teachers in intervention schools were trained to deliver health lessons and to refer sick students to care. This study is designed as a prospective matched control study. Students from the seven intervention schools are matched with students from control schools.

ELIGIBILITY:
Inclusion Criteria:

* Children attending one of the 14 schools in the study.

Exclusion Criteria:

* Children not attending one of the 14 schools in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of acute disease | Baseline, 6 months, and one-year follow-up
  Students report on the presence of 14 systemic, genitourinary, respiratory, and gastrointestinal illnesses in the past two week. Acute illnesses are combined into a summary index of morbidity.

SECONDARY OUTCOMES:
Change in weight | Baseline, 6 months, and one-year follow-up
  Calculate body mass index (BMI)-for-age z-scores using the World Health Organization AnthroPlus Software macro for Stata. Thinness and overweightness are defined respectively as: BMI-for-age below -2 SD and as BMI-for-age above 1 standard deviation.
Change in height | Baseline, 6 months, and one-year follow-up
  Calculate standardized height-for-age (HAZ) z-scores using the World Health Organization AnthroPlus Software macro for Stata. Stunting was defined as HAZ below -2 standard deviation.
Change in health knowledge | Baseline, 6 months, and one-year follow-up
  Calculate the percentage of correct answers on 11-question quiz on various health topics.
Change in school attendance | Baseline, 6 months, and one-year follow-up
  Calculate percentage of students who missed one or more days from school in the past two weeks.
Change in academic performance | Baseline, 6 months, and one-year follow-up
  Students report on their own school performance and academic performance is verified by term marks.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei D, Brigell R, Khadka A, Perales N, Fink G. Comprehensive school-based health programs to improve child and adolescent health: Evidence from Zambia. PLoS One. 2019 May 31;14(5):e0217893. doi: 10.1371/journal.pone.0217893. eCollection 2019. PMID 31150484